CLINICAL TRIAL: NCT00515567
Title: Utilization of Explanted Lungs for Isolation of Tissue Samples and Primary Cell Lines to Study Pulmonary Fibrosis
Brief Title: Explanted Lung Tissues With Pulmonary Fibrosis
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 14514A
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Fibrosis
Keywords: explanted lungs; pulmonary fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — explanted lung tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to use the tissues from the explanted lungs in order to better study the cause of pulmonary fibrosis at a cellular level.

DETAILED DESCRIPTION:
Pulmonary Fibrosis involves scarring of the lung. Gradually, the air sacs of the lungs become replaced by fibrotic tissue. The most current thinking is that the fibrotic process is a reaction to tiny injury to the lung. When the scar forms, the tissue becomes thicker causing a permanent loss of the tissue's ability to carry oxygen into the bloodstream.

We need to obtain lung tissue from patients without pulmonary fibrosis and compare it to lung tissue from patients with pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* all patients awaiting lung transplant

Exclusion Criteria:

* all who will not give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects listed for lung transplant
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2006-02; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
assess fibroblasts and cytokines associated with pulmonary fibrosis | 12/2013

CONTACTS AND LOCATIONS:
Overall Officials: Nickolai Dulin, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States